CLINICAL TRIAL: NCT06885437
Title: Neonatal Intensive Care Nurses' Assessment of Preterm Infants' Pain and Sedation: Inter-Rater Reliability
Brief Title: Neonatal Intensive Care Nurses' Assessment of Preterm Infants' Pain and Sedation
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Other Study IDs: ATADEK-2022-20/25
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Nurse Care Coordination
Keywords: preterm; nurse; pain; N-PASS
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preterm infant: Preterm infants undergoing pain and sedation assessment by NICU nurses
  Interventions: Other: Pain and sedation assessment with the N-PASS scale by each nurse

INTERVENTIONS:
Other: Pain and sedation assessment with the N-PASS scale by each nurse — After a painful procedure, the infant's N-PASS pain and sedation scores were assessed simultaneously by three observers (two researchers and the patients' head nurses) independently and blinded.

SUMMARY:
The aim of this study was to investigate the consistency of NICU nurses' assessment of pain and sedation using NPASS in preterm infants in the NICU

DETAILED DESCRIPTION:
The experience of pain is a common occurrence for infants in NICUs, with many undergoing painful procedures for diagnostic or therapeutic purposes. Effective pain management is a critical issue, as repeated painful experiences and stress in the early stages of life have the potential to have adverse short- and long-term effects on infant health. Although the importance of assessment and management of pain in neonates is well known, these practices still need to be improved in the NICU. Firstly, pain and sedation assessment with reliable tools is needed to provide adequate pain management practices. Because the evaluation of the pain and sedation level directs the treatment, thus avoiding inadequate or unnecessary treatment applied to the infants. However, the assessment of pain in newborns is a challenging endeavor, due to the inability of this age group to communicate, the existence of variations in pain responses based on age, the lack of training in the recognition of pain in premature infants, and the practical limitations of current assessment tools. Therefore, this study aimed to assess the inter-rater reliability of the N-PASS in a clinical actual setting. In this context, there needs to be consistency between assessors in pain assessment. As a result, the aim of this study was to investigate the consistency of NICU nurses' assessment of pain and sedation using NPASS in preterm infants in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in the NICU for at least six months and agreeing to participate in the study
* Preterm infant

Exclusion Criteria:

* Less than six months of NICU experience
* Term infant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses with more than 6 months of experience working in the neonatal intensive care unit and preterm newborns cared by these nurses constitute the population.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
N-PASS score observed by different nurses at the same time | NPASS score will be assessed once daily for 10 days by different nurses at the same time
  The N-PASS scores were assigned by three observers (two researchers and nurses).Each patient's primary nurse and the two researchers were given 1 minute to independently record the patient's total N-PASS score. Observers recorded post-assessment pain and sedation scores separately after each assessment. The nurses and two researchers remained blind to each other's evaluations and submitted the forms they filled out individually.The N-PASS, , includes four behavioral items (crying irritability, behavior state, facial expression, extremities tone) and one vital signs item (changes in heart rate, respiratory rate, blood pressure, and oxygen saturation). Each pain criterion is scored on a scale of 0, 1 and 2. The maximum score on the N-PASS is 11 for preterm infants under 30 weeks and 10 for preterm infants over 30 weeks. Pain intensity is categorized as no pain (0-3), mild pain (4-7) and severe pain (8-11).

CONTACTS AND LOCATIONS:
Overall Officials: Selvinaz Albayrak, Assist. Prof., Principal Investigator — Istinye University
Locations (1):
- Acıbadem University, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llerena A, Tran K, Choudhary D, Hausmann J, Goldgof D, Sun Y, Prescott SM. Neonatal pain assessment: Do we have the right tools? Front Pediatr. 2023 Feb 2;10:1022751. doi: 10.3389/fped.2022.1022751. eCollection 2022. PMID 36819198
- [Background] Pavlyshyn H, Sarapuk I, Kozak K. The relationship between neonatal stress in preterm infants and developmental outcomes at the corrected age of 24-30 months. Front Psychol. 2024 May 22;15:1415054. doi: 10.3389/fpsyg.2024.1415054. eCollection 2024. PMID 38840740
- [Background] Luo F, Zhu H, Mei L, Shu Q, Cheng X, Chen X, Zhao Y, Chen S, Pan Y. Evaluation of procedural pain for neonates in a neonatal intensive care unit: a single-centre study. BMJ Paediatr Open. 2023 Oct;7(1):e002107. doi: 10.1136/bmjpo-2023-002107. PMID 37821124
- [Background] Campbell-Yeo M, Eriksson M, Benoit B. Assessment and Management of Pain in Preterm Infants: A Practice Update. Children (Basel). 2022 Feb 11;9(2):244. doi: 10.3390/children9020244. PMID 35204964